CLINICAL TRIAL: NCT06417307
Title: Supervised Exercise Therapy on Mitochondrial Functions of Platelet and Lymphocyte in Patients With End-Stage Renal Disease on Hemodialysis
Brief Title: Exercise on Mitochondrial Functions of Lymphocyte in Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, Consultant, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202002321A3C501
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-05

CONDITIONS: Hemodialysis Complication
Keywords: Hemodialysis; Mitochondria; Lymphocyte; Exercise training
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervised exercise training (Experimental): Moderate intensity continuous cycling training.
  Interventions: Behavioral: Supervised exercise training
- Control group (Experimental): Recieve no intervention but only maintain daily lifestyle.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Supervised exercise training — Participants perform Intradialytic cycling exercise training in the hospital for 6 months (24 weeks) and 3 months (12 weeks) at home. Exercise prescription: 50-60% maximal workload for 20-30 minutes, including low intensity warm-up and cool down (30% of maximal workload).
  Arms: Supervised exercise training
Behavioral: Control group — Maintain daily lifestyle until the end of the study. Receive no intervention/supplements.
  Arms: Control group

SUMMARY:
To improve aerobic capacity, muscular function and health-related quality of life in patients with end-stage renal disease (ESRD), regular exercise is recommended. Supervised intradialytic exercise with moderate intensity is an available approach to maintain patients' safety and compliance, and enhance physiological adaptations effectively. The exercise training effects of mitochondrial functions of lymphocyte in ESRD patients, like respiratory capacity, bioenergetic status and thrombosis/immunological regulation remained unclear.

Method: ESRD patients (anticipated n=180) would conduct supervised exercise training therapy for 3 days a week for 6 months in the hospital and 3 months at home. Cardiopulmonary exercise therapy would be performed before and after the intervention. A high resolution respirometer and a flow cytometer are used to determine the oxygen consumption rate/mitochondrial respiration in mitochondria and subtypes of lymphocyte, respectively.

DETAILED DESCRIPTION:
Renal dysfunction results from cardiovascular-related comorbidities or metabolic disorders, accumulating excessive inflammatory products or damage mitochondrial bioenergetics health in platelet and lymphocyte, then lead to chronic kidney disease (CKD) eventually. End-stage renal disease (ESRD) is the highest level of CKD, patients at ESRD stage suffer from severe uremia and renal failure, preparing renal replacement therapy: dialysis.

Hemodialysis (HD) are the most common treatment for ESRD patients, especially in Taiwan, where reports the highest prevalence of HD globally due to related chronic diseases and comprehensive National Health Insurance program. Maintenance (long-term) HD results in physical inactivity and low quality of life; thus, exercise training is recommended to improve physiological adaptations and functional capacity for HD patients. With supervised condition and a safer progression, intradialytic exercise in clinical settings provides low dropout rate and superior compliance.

Mitochondrial dysfunction is one of the concerned issues in ESRD, impaired mitochondria also dysregulate circulating lymphocyte, leading to immunological senescence .

The purposes of the present study are to establish the measurements of mitochondrial functions of platelet and lymphocyte in HD patients, and determine cardiovascular and muscular fitness along with the effects of intradialytic exercise.

ELIGIBILITY:
Inclusion Criteria:

* All patients have been receiving hemodialysis and medication at least for 6 weeks, the Kt/V score must be above 1.2 to show that they were stable.

Exclusion Criteria:

* Under 20 years-old, hyperkalemia occurs within 3 month, orthopedic or muscular diseases, other medical, psychological or physiological diseases, pregnancy exercise contraindications.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Mitochondrial function of lymphocyte | 9 months
  Evaluate oxygen consumption rate (oxidative phophorylation/electron transport chain), bioenergetic health index (BHI) in lymphocyte by using a high resolution respirometer.
  Evaluate mitochondrial function and subtypes of lymphocyte by using a aflow cytometer.

SECONDARY OUTCOMES:
Cardiopulmonary fitness | 9 months
  ESRD patients performed cardiopulmonary exercise testing (CPET) to assess their aerobic capacity. CPET composed of continuous workload increment of 10 W/min until exhaustion (usually within 8-12 minutes). Oxygen consumption, carbon dioxide production, ventilation, respiratory rate would be recorded.
Quality of life in ESRD patients | 9 months
  We would use a qusionnaire named ESRDkidney disease quality of life-36 (KDQOL-36) to record and scale the qulaity of life in ESRD patients. The content include work status, cognitive funtion, social support, physical functioning and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Shyan Wang, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung University, Taoyuan District, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altintas MM, DiBartolo S, Tadros L, Samelko B, Wasse H. Metabolic Changes in Peripheral Blood Mononuclear Cells Isolated From Patients With End Stage Renal Disease. Front Endocrinol (Lausanne). 2021 Mar 9;12:629239. doi: 10.3389/fendo.2021.629239. eCollection 2021. PMID 33790861
- [Background] Deligiannis A, D'Alessandro C, Cupisti A. Exercise training in dialysis patients: impact on cardiovascular and skeletal muscle health. Clin Kidney J. 2021 Jan 11;14(Suppl 2):ii25-ii33. doi: 10.1093/ckj/sfaa273. eCollection 2021 Apr. PMID 33981417
- [Background] Chou CH, Fu TC, Tsai HH, Hsu CC, Wang CH, Wang JS. High-intensity interval training enhances mitochondrial bioenergetics of platelets in patients with heart failure. Int J Cardiol. 2019 Jan 1;274:214-220. doi: 10.1016/j.ijcard.2018.07.104. Epub 2018 Jul 27. PMID 30072155
- [Background] Lopes LCC, Mota JF, Prestes J, Schincaglia RM, Silva DM, Queiroz NP, Freitas ATVS, Lira FS, Peixoto MDRG. Intradialytic Resistance Training Improves Functional Capacity and Lean Mass Gain in Individuals on Hemodialysis: A Randomized Pilot Trial. Arch Phys Med Rehabil. 2019 Nov;100(11):2151-2158. doi: 10.1016/j.apmr.2019.06.006. Epub 2019 Jul 3. PMID 31278924
- [Background] Sovatzidis A, Chatzinikolaou A, Fatouros IG, Panagoutsos S, Draganidis D, Nikolaidou E, Avloniti A, Michailidis Y, Mantzouridis I, Batrakoulis A, Pasadakis P, Vargemezis V. Intradialytic Cardiovascular Exercise Training Alters Redox Status, Reduces Inflammation and Improves Physical Performance in Patients with Chronic Kidney Disease. Antioxidants (Basel). 2020 Sep 15;9(9):868. doi: 10.3390/antiox9090868. PMID 32942555